CLINICAL TRIAL: NCT06968689
Title: Spatiotemporal Thalamocortical Alterations Underlie Experimental and Chronic Pain - Phase II
Brief Title: Spatiotemporal Thalamocortical Alterations Underlie Experimental and Chronic Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Wen Li, Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: HSC-MS-25-0062; 5R01NS129059-03 (NIH)
Record Dates: First submitted 2025-05-05; First posted 2025-05-13 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2025-05

CONDITIONS: Pain
Keywords: Transcranial Alternating Current Stimulation (tACS)
MeSH Terms: conditions — Pain | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (6):
- tACS then tRNS then sham (Experimental)
  Interventions: Device: transcranial alternating current stimulation (tACS); Device: Sham; Device: transcranial random noise stimulation (tRNS)
- tACS then sham then tRNS (Experimental)
  Interventions: Device: transcranial alternating current stimulation (tACS); Device: Sham; Device: transcranial random noise stimulation (tRNS)
- tRNS then tACS then sham (Experimental)
  Interventions: Device: transcranial alternating current stimulation (tACS); Device: Sham; Device: transcranial random noise stimulation (tRNS)
- tRNS then sham then tACS (Experimental)
  Interventions: Device: transcranial alternating current stimulation (tACS); Device: Sham; Device: transcranial random noise stimulation (tRNS)
- Sham then tRNS then tACS (Experimental)
  Interventions: Device: transcranial alternating current stimulation (tACS); Device: Sham; Device: transcranial random noise stimulation (tRNS)
- Sham then tACS then tRNS (Experimental)
  Interventions: Device: transcranial alternating current stimulation (tACS); Device: Sham; Device: transcranial random noise stimulation (tRNS)

INTERVENTIONS:
Device: transcranial alternating current stimulation (tACS) — Participants will get a personalized brain stimulation: a 2 milliampere (mA) oscillating current that matches their natural alpha brain wave frequency (8-12 Hz), determined by a quick 3-minute EEG before the session.
Device: Sham — Active sham stimulation with 60- second -tACS will be applied , then ramp down, and be reintroduced in the last 30 seconds to minimize awareness of the experimental condition
Device: transcranial random noise stimulation (tRNS) — Participants will still get stimulation, but at random frequencies between 1 and 200 Hz (instead of targeted alpha waves).

SUMMARY:
The purpose of this study is to assess thalamocortical (TC) connectivity during tonic pressure pain, to evaluate alpha activity during tonic pressure pain and to determine pressure pain ratings by using Electroencephalography (EEG), Functional Magnetic Resonance Imaging (fMRI), Transcranial Alternating Current Stimulation (tACS), sham and Transcranial random noise stimulation (tRNS)

ELIGIBILITY:
Inclusion Criteria:

* Meet the MRI / EEG screening criteria
* Fluent in English

Exclusion Criteria:

* Current or history of major medical, neurological, or psychiatric illness based on self-report
* History of cardiac, respiratory, or nervous system disease that, in the investigator's judgment, precludes participation in the study because of a heightened potential for adverse outcome (for example: asthma or claustrophobia)
* History of head trauma
* Pregnant or lactating
* Presence of any contraindications to MRI scanning (for example: cardiac pacemaker, metal implants, claustrophobia, pregnancy, cannot lie still in fMRI scanner)
* Conditions making study participation difficult (e.g., paralysis, psychoses, or other severe psychological problems as per the judgment of a study investigator during Session 1)
* Active substance abuse disorders (based on subject self-report)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-05-12 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in thalamocortical (TC) connectivity during tonic pressure pain using fMRI | pre-stimulation, post-stimulation (about 30 minutes)
Change in alpha activity during tonic pressure pain using EEG | pre-stimulation, post-stimulation (about 30 minutes)

SECONDARY OUTCOMES:
Change in pain as assessed by the Visual Analog Scale (VAS) | pre-stimulation, post-stimulation (about 30 minutes)
  The VAS is scored from 0 = no pain; 10 = the most intense pain tolerable, higher number indicating more pain

CONTACTS AND LOCATIONS:
Overall Officials: Wen Li, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No